CLINICAL TRIAL: NCT01660581
Title: A Randomized,Prospective,Double-blind Study to Evaluate Intracardiac Injections of Bone Marrow,Autologous CD133+Cells(Electromechanical Mapping Based)in Patients With Resistant Angina and no Effective Revascularization Option. RegentVsel
Brief Title: Intracardiac CD133+ Cells in Patients With No-option Resistant Angina
Acronym: RegentVsel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Wojciech Wojakowski MD, PhD, MD, PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Regent Vsel; 2011-005435-98 (EudraCT Number)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Stable Angina
Keywords: CD133+; stem cells; Coronary Artery Disease; Stable Angina Pectoris
MeSH Terms: conditions — Angina, Stable; Macular Dystrophy, Retinal, 2; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD133+ (Experimental): intramyocardial injection (electromechanical mapping based) of autological CD133+ cells, isolated from bone marrow
  Interventions: Biological: intramyocardial injection (electromechanical mapping based)
- Placebo (Placebo Comparator): intramyocardial injection (electromechanical mapping based) of placebo - 0,9% NaCl plus 0,5% solution of patients' serum
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: intramyocardial injection (electromechanical mapping based) — Patient will undergo 3D electric and mechanical intracardiac mapping; based on maps generated intramyocardial administration of autologous CD133+ cells or placebo will be performed.
  Arms: CD133+
Biological: Placebo — Patients in the placebo group receive 0.9% NaCl solution with 0.5% solution of the patient's own serum.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of therapy with autological CD133+ cells in patients with angina resistant to pharmacological treatment and without the possibility of effective revascularization. Cells will be isolated from patients bone marrow and administered directly into the muscle of left ventricle. The main objective is to assess the treatments' influence on improvement of myocardial perfusion and function, and on decrease of occurrence of symptomatic angina.

DETAILED DESCRIPTION:
Patients with a Stable angina pectoris (CCS II-IV) can potentially benefit from treatment with autological CD133+ cell populations, which include cells with a higher expression of cardiac and endothelial differentiation markers.

REGENT VSEL Trial will include Patients with Angina resistant to pharmacological treatment and without the possibility of effective revascularization.

The main objective of the study is to assess the treatments influence on:

* improvement of myocardial perfusion
* global and segmental contractility (LVEF)
* occurrence of symptomatic angina
* quality of life

Regent Vsel is a prospective, randomized, double blind, placebo-controlled study with a planned number of 60 Patients.

Randomization will be carried out according to a 1:1 mode. Every Patient will undergo a bone marrow aspiration. CD133+ cells will be isolated from bone marrow aspirates. Patients randomized to experimental group will receive isolated cells (direct left ventricular muscle administration). Patients enrolled to control group will get only a placebo solution injected into the muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Stable angina CCS II-IV despite maximum pharmacotherapy for at least 2 weeks since last medications change
2. Presence of ≥ 1 myocardial segment with ischemia features in Tc-99m SPECT
3. Patients disqualified from revascularization procedures by Heart Team
4. Patient age > 18 and < 75 year old
5. Patient must provide written informed consent for participation in study

Exclusion Criteria:

1. Acute coronary syndrome in less than 6 months prior to enrollment
2. Heart failure NYHA III-IV
3. LVEF <35%
4. Presence of intracardiac thrombus (echocardiography confirmed), massive calcification of the aortic valve and left ventricular aneurysm
5. Previous cardioverter-defibrillator or cardiac stimulator implantation
6. Allergy to contrast agents
7. History of malignancy
8. HIV, HBV, HCV infection
9. Life expectancy less than 6 months
10. Bleeding diathesis
11. Renal insufficiency (GFR < 30 mL/min/1.73m2)
12. Pregnancy, lactation, or ineffective contraception in women of childbearing potential

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion change | 4 months after application of cell therapy
  Myocardial perfusion change assessed by perfusion scintigraphy (99mTc SPECT)

SECONDARY OUTCOMES:
Global and segmental contractility change and myocardial perfusion change | MRI 4 months and echocardiography 4 and 12 months after application of cell therapy
  Global and segmental contractility change and myocardial perfusion change assessed by magnetic resonance imaging with adenosine administration, and echocardiography with contrast
Exercise tolerance | 4 and 12 months after application of cell therapy
  Exercise tolerance assessed in a treadmill test (TET, ESTD, TTLA)
Occurrence of symptomatic angina | 1, 4, 6 and 12 months after application of cell therapy
  CCS, nitrates usage
Quality of life | 1, 4, 6 and 12 months after application of cell therapy
  Quality of life assessed by standard questionnaires: SF37, Seattle Angina
Occurrence of ventricular arrhythmia | 1, 4, 6 and 12 months after application of cell therapy
  24 hrs ECG monitoring
Occurrence of in-stent restenosis and progression of artherosclerotic lesions in remained coronary artery segments | 4 months after application of cell therapy
  Assessed by Intravascular Ultrasound (IVUS) and Optical coherence tomography (OCT) examination

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Wojakowski, MD, PhD, Principal Investigator — Samodzielny Publiczny Szpital Kliniczny nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach Górnośląskie Centrum Medyczne III Klinika Kardiologii
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach Górnośląskie Centrum Medyczne im. prof. Leszka Gieca, Katowice-Ochojec, Silesian, Poland

REFERENCES:
- [Background] Abdel-Latif A, Bolli R, Tleyjeh IM, Montori VM, Perin EC, Hornung CA, Zuba-Surma EK, Al-Mallah M, Dawn B. Adult bone marrow-derived cells for cardiac repair: a systematic review and meta-analysis. Arch Intern Med. 2007 May 28;167(10):989-97. doi: 10.1001/archinte.167.10.989. PMID 17533201
- [Background] Lipinski MJ, Biondi-Zoccai GG, Abbate A, Khianey R, Sheiban I, Bartunek J, Vanderheyden M, Kim HS, Kang HJ, Strauer BE, Vetrovec GW. Impact of intracoronary cell therapy on left ventricular function in the setting of acute myocardial infarction: a collaborative systematic review and meta-analysis of controlled clinical trials. J Am Coll Cardiol. 2007 Oct 30;50(18):1761-7. doi: 10.1016/j.jacc.2007.07.041. Epub 2007 Oct 15. PMID 17964040
- [Background] Wojakowski W, Tendera M, Zebzda A, Michalowska A, Majka M, Kucia M, Maslankiewicz K, Wyderka R, Krol M, Ochala A, Kozakiewicz K, Ratajczak MZ. Mobilization of CD34(+), CD117(+), CXCR4(+), c-met(+) stem cells is correlated with left ventricular ejection fraction and plasma NT-proBNP levels in patients with acute myocardial infarction. Eur Heart J. 2006 Feb;27(3):283-9. doi: 10.1093/eurheartj/ehi628. Epub 2005 Nov 2. PMID 16267071
- [Background] Wojakowski W, Tendera M, Michalowska A, Majka M, Kucia M, Maslankiewicz K, Wyderka R, Ochala A, Ratajczak MZ. Mobilization of CD34/CXCR4+, CD34/CD117+, c-met+ stem cells, and mononuclear cells expressing early cardiac, muscle, and endothelial markers into peripheral blood in patients with acute myocardial infarction. Circulation. 2004 Nov 16;110(20):3213-20. doi: 10.1161/01.CIR.0000147609.39780.02. Epub 2004 Nov 8. PMID 15533859
- [Background] van Ramshorst J, Bax JJ, Beeres SL, Dibbets-Schneider P, Roes SD, Stokkel MP, de Roos A, Fibbe WE, Zwaginga JJ, Boersma E, Schalij MJ, Atsma DE. Intramyocardial bone marrow cell injection for chronic myocardial ischemia: a randomized controlled trial. JAMA. 2009 May 20;301(19):1997-2004. doi: 10.1001/jama.2009.685. PMID 19454638
- [Background] Dimmeler S, Burchfield J, Zeiher AM. Cell-based therapy of myocardial infarction. Arterioscler Thromb Vasc Biol. 2008 Feb;28(2):208-16. doi: 10.1161/ATVBAHA.107.155317. Epub 2007 Oct 19. PMID 17951319
- [Derived] Wojakowski W, Jadczyk T, Michalewska-Wludarczyk A, Parma Z, Markiewicz M, Rychlik W, Kostkiewicz M, Gruszczynska K, Blach A, Dzier Zak-Mietla M, Wanha W, Ciosek J, Ochala B, Rzeszutko L, Cybulski W, Partyka L, Zasada W, Wludarczyk W, Dworowy S, Kuczmik W, Smolka G, Pawlowski T, Ochala A, Tendera M. Effects of Transendocardial Delivery of Bone Marrow-Derived CD133+ Cells on Left Ventricle Perfusion and Function in Patients With Refractory Angina: Final Results of Randomized, Double-Blinded, Placebo-Controlled REGENT-VSEL Trial. Circ Res. 2017 Feb 17;120(4):670-680. doi: 10.1161/CIRCRESAHA.116.309009. Epub 2016 Nov 30. PMID 27903568